CLINICAL TRIAL: NCT00163878
Title: A Randomised Control Trial to Determine the Effectiveness of Sensory Stimulation Program in Reducing the Length of Time Spent by Severely Brain Injured Patients in a Vegetative State in the Acute Hospital Environment
Brief Title: Is Sensory Stimulation Effective in Reducing Time Spent in a Coma or Vegetative State
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Victorian Trauma Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4468
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2005-08

CONDITIONS: Traumatic Brain Injury
Keywords: Sensory Stimulation Programs
MeSH Terms: conditions — Brain Injuries, Traumatic

INTERVENTIONS:
Procedure: Sensory Stimulation
Device: Sesnory Modality Assessment and Rehabilitation Technique

SUMMARY:
A randomised control trial of patients who have a severe brain injury to determine if patients who receive a standardised sensory stimulation program emerge earlier from a vegetative state. The experimental group would receive, in addition to their normal occuaptional therapy, sensory stimulation which would involve the daily application of stimulation to all five senses using the Sensory Modalities Assessment and Rehabilitation Technique (SMART).

DETAILED DESCRIPTION:
A randomised control trial of patients who have a severe brain injury to determine if patients who receive a standardised sensory stimulation program emerge earlier from a vegetative state. The experimental group would receive, in addition to their normal occupational therapy, sensory stimulation which would involve the daily application of stimulation to all five senses using the Sensory Modalities Assessment and Rehabilitation Technique (SMART).

The SMART is both an assessment and treatment too. Patients in both groups will have baseline assessments conducted using the SMART, with further assessments conducted every ten days for thrity days. The SMART is designed to provide quantitative data in the assessment of the patients cognitive function and potential awareness. It is a five point hierarchical scale from level 1 ( no response) to level 5 (discriminating).

ELIGIBILITY:
Inclusion Criteria:

* admitted with severe brain injury
* GCS of 9 or less. A GCS score of 9 or less is indicative of a severe brain injury
* medically stable, as documented by medical staff
* age 18 to 65 years
* controlled intracranial pressure no sedation
* no previous brain injury

Exclusion Criteria

* patient declared brain dead
* next of kin withdraws patient from the study
* withdrawal of consent by patient on waking
* raised uncontrolled intracranial pressure, following discussions with treating medical team
* patient enrolled in DECRA or RSI Trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Study Completion 2006-12

PRIMARY OUTCOMES:
Patients are allocated to a level on the SMART scale every ten days, compariosns are made between the control and experimental groups

SECONDARY OUTCOMES:
Fucntional status at six months, assessed using the modified Barthel

CONTACTS AND LOCATIONS:
Overall Officials: Jacqui M Morarty, Occupational Therapist, Principal Investigator — Bayside Health
Locations (2):
- Australia (2):
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - The Alfred Hosptial, Melbourne, Victoria